CLINICAL TRIAL: NCT03090581
Title: Prospective Study of Transbronchial Biopsies With Cryoprobe in Patients With Lung Transplantation Admitted to an Intensive Care Unit.
Brief Title: Transbronchial Biopsies With Cryoprobe in Patients With Lung Transplantation.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CB JKMT-1
Record Dates: First submitted 2017-03-08; First posted 2017-03-27 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Lung Transplant Rejection
Keywords: Graft Rejection/diagnosis; Lung Transplantation; Cryoprobe
MeSH Terms: conditions — Disease

STUDY DESIGN:
Masking Description: A prospective, randomized, comparative study in all patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Biopsies CP 1 (Active Comparator): Obtain transbronchial lung biopsies with cryoprobe (CP) 1
  Interventions: Procedure: Biopsies CP
- Biopsies CP 2 (Active Comparator): Obtain transbronchial lung biopsies with cryoprobe (CP) 2
  Interventions: Procedure: Biopsies CP
- Biopsies FC (Active Comparator): Obtain transbronchial lung biopsies with forceps (FC).
  Interventions: Procedure: Biopsies FC

INTERVENTIONS:
Procedure: Biopsies CP — Transbronchial biopsies will be obtained with a flexible bronchoscope, using a cryoprobe.
  Arms: Biopsies CP 1; Biopsies CP 2
Procedure: Biopsies FC — Transbronchial biopsies will be obtained with a flexible bronchoscope, using a forceps.
  Arms: Biopsies FC

SUMMARY:
The survival of lung transplant patients (PD) is limited mainly by Infections, graft dysfunction in the immediate postoperative period and chronic dysfunction. Up to 36% have an episode of acute rejection after transplantation. For the diagnosis of these pathologies, transbronchial lung biopsy (BPTB) is essential. The classical method is the realization of BPTB with conventional clamp, but the performance diagnosis is limited. However, the use of cryoprobes for sampling in other pulmonary pathologies have been shown to achieve a higher diagnostic yield. The BPTB performance is variable and depends on factors such as sample size and the presence of artifacts (crushing) produced by the forceps tweezers. The objective principal is to compare the diagnostic yield of samples obtained with cryoprobe compared to those obtained with conventional biopsy tweezers. A prospective, randomized, and comparative study is proposed for all patients in the intensive care unit after lung transplantation in a 24-month period, at Vall de Hebron Hospital. Patients will be divided into two groups: symptomatic and asymptomatic. The exclusion criteria are the contraindications of the procedure and the factors which increase the hemorrhagic risk. A flexible bronchoscope (BF-18BS) will be used and the procedure will be performed according to the technique conventional. The patient undergoing the procedure will be intubated, sedated and relaxed under supervision and continuous monitoring by an intensivist. A bronchoalveolar lavage and a maximum of 6 samples will be obtained. Morphological study (middle area, artifacts, components, diagnosis), microbiological, histological and anatomopathological according to the usual protocol. The duration of the procedure, the complications and the frequency with which the diagnosis obtained after the procedure modifies the therapeutic behavior will be monitored. These data will allow to evaluate the potential benefits of this procedure in the diagnosis of pulmonary pathology in lung transplantation.

DETAILED DESCRIPTION:
Bronchoscopic examinations will be performed with intubated patients under continuous monitoring (pulse oximetry, blood pressure, heart and respiratory rate), Oxygen therapy with high flows and surveillance by anesthesiologist. The bronchopulmonary lobe where the biopsies will be performed is determined prior to the procedure based on an imaging study (chest x-ray or computed tomography). Transbronchial biopsies will be obtained using a flexible bronchoscope (Pentax, 3.2 mm working channel), which approaches the subsegment where the affected area is located. The 2.4 mm diameter cryoprobe is placed (Erbokryo®), and moves forward until it encounters a soft resistance. The cryoprobe is removed between 5-10 mm and the freezing is applied for 3 seconds. After 3 seconds, the probe is gently removed together with the bronchoscope and frozen tissue sample at the tip of the probe. In the case of strong resistance, the process is stopped and then repeated. In the case of the use of forceps, the conventional technique is used.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary transplant patients admitted to the intensive care unit who are assigned a transbronchial lung biopsy.

Exclusion Criteria:

* Respiratory insufficiency refractory to oxygen therapy.
* Acute or subacute ischemic heart disease.
* Severe arrhythmias.
* Coagulation disorders: platelets < 60,000-50,000 or Prothrombin time > 60%.
* Lack of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2017-03-15 (Actual); Primary Completion 2018-01 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Number of patients in whom a pathological diagnosis is obtained after obtaining transbronchial biopsies, performed with forceps or cryosondes. | 5 days after biopsies
  Graft rejection is classified according to the criteria of the International Society for Heart and Lung Transplantation (ISHLT) in 2007.

SECONDARY OUTCOMES:
Number of alveoli, bronchioles, bronchi, blood vessels and pleura containing each biopsy. | 5 days after biopsies
  A microscope will be used with Software Mese. ¨Leica Application Suite X¨.
Number of complications related to the procedure. | 30 days after biopsies
  Complications: bleeding, pneumothorax, infection or acute respiratory failure.

CONTACTS AND LOCATIONS:
Overall Officials: Javier De Gracia, Pneumologist, Principal Investigator — Respiratory department; Karina I Loor, MD, Study Chair — Respiratory department; Mario Culebras, MD, Study Chair — Respiratory department; Antonio Álvarez, MD, Study Chair — Respiratory department
Locations (1):
- Hospital Vall de Hebron., Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No
no.

REFERENCES:
- [Derived] Loor K, Culebras M, Sansano I, Alvarez A, Sacanell J, Garcia-de-Acilu M, Berastegui C, Polverino E, Clofent D, de Gracia J. Lung allograft transbronchial cryobiopsy for critical ventilated patients: a randomised trial. Eur Respir J. 2023 Jan 6;61(1):2102354. doi: 10.1183/13993003.02354-2021. Print 2023 Jan. PMID 35896217